CLINICAL TRIAL: NCT04286035
Title: Comparison of the Effects of Femoral Nerve Block and Adductor Canal Block on Postoperative Analgesia in Patients Undergoing Unilateral Total Knee Arthroplasty
Brief Title: Two Different Blocks for Postoperative Analgesia in Patients Undergoing Unilateral Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kerim Şahin, Research assistant, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SK01
Record Dates: First submitted 2020-02-21; First posted 2020-02-26 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Knee Replacement, Total; Pain, Postoperative; Anesthesia, Regional
Keywords: femoral nerve block, adductor canal block, total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral group (Active Comparator)
  Interventions: Drug: Bupivacaine Injection
- Adductor group (Active Comparator)
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Bupivacaine Injection — Femoral nerve block with 20 ml %0.375 bupivacaine
  Arms: Femoral group
Drug: Bupivacaine Injection — Adductor canal block with 20 ml %0.375 bupivacaine
  Arms: Adductor group

SUMMARY:
The frequency of femoral nerve block and adductor canal block for analgesia after TKA(total knee arthroplasty) increases with the use of ultrasonography in regional anesthesia. In this study, we aimed to compare the effects of femoral nerve block and adductor canal block on postoperative analgesia in patients undergoing unilateral knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* ASA(American Society of Anesthesiologists) Classification I-II
* Age: <55 years
* Unilateral total knee arthroplasty

Exclusion Criteria:

* Does not approve the study
* Pregnant
* Emergency
* ASA III-IV
* History of local anesthetic allergy
* Infection in the block area
* Coagulation disorder
* Morbid obesity (body mass index> 40 kg / m²)
* Severe organ failure
* Previous neurological deficit
* Psychiatric disease
* History of chronic pain

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Tramadol consumption | 24 hours after operation
  Postoperative tramadol consumption with patient controlled analgesia
VAS(visual analogue scale) score (0-10, 0 is no pain, 10 is the most severe pain) | 24 hours after operation
  VAS(visual analogue scale) score (0-10, 0 is no pain, 10 is the most severe pain) is less than four is adequate analgesia
Rescue analgesic requirement | 24 hours after operation
  If VAS(visual analogue scale) score (0-10, 0 is no pain, 10 is the most severe pain) is is four or more, paracetamol 1000 mg is administered

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | 24 hours after operation
  Frequency of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Şişli Hamidiye Etfal Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No